CLINICAL TRIAL: NCT05809895
Title: AdvanTIG-211: A Randomized, Double-blind, Placebo-controlled, Phase II Study Evaluating the Efficacy and Safety of Ociperlimab (WCD118) Combined With Tislelizumab (VDT482) Plus Chemotherapy Versus Placebo Combined With Pembrolizumab Plus Chemotherapy as First-line Therapy for Participants With Advanced Triple Negative Breast Cancer (TNBC)
Brief Title: Phase II Study Evaluating the Efficacy and Safety of Ociperlimab in Combination With Tislelizumab and Chemotherapy as First-line Treatment for Participants With Advanced Triple Negative Breast Cancer
Acronym: AdvanTIG-211
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision, not driven by safety concerns; no new safety signals have been observed in the ociperlimab program.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CWCD118B12201; 2022-503099-99-00 (Other: EU CTIS number)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; Triple Negative Breast Cancer; PD-L1; Ociperlimab; Tislelizumab; WCD118 (BGB-A1217); VDT482 (BGB-A317); Pembrolizumab; Carboplatin; Gemcitabine; Paclitaxel; Nab-paclitaxel; TIGIT; Combination immunotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — tislelizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Carboplatin; pembrolizumab; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized to Arms A, B and C in a double-blind manner Participants will be enrolled in Arm D in an open-label manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: ociperlimab+tislelizumab+chemotherapy (PD-L1 CPS ≥ 10) (Experimental): Participants with a PD-L1 CPS ≥ 10 will receive after randomization ociperlimab + tislelizumab + chemotherapy. The choice of one of three chemotherapy options is at the discretion of the investigator provided that it is either: (1) paclitaxel, (2) nab-paclitaxel, or (3) gemcitabine plus carboplatin.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Gemcitabine
- Arm B: placebo + pembrolizumab + chemotherapy (PD-L1 CPS ≥ 10) (Active Comparator): Participants with a PD-L1 CPS ≥ 10 will receive after randomization placebo + pembrolizumab + chemotherapy. The choice of one of three chemotherapy options is at the discretion of the investigator provided that it is either: (1) paclitaxel, (2) nab-paclitaxel, or (3) gemcitabine plus carboplatin.
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Placebo; Drug: Pembrolizumab; Drug: Gemcitabine
- Arm C: placebo + tislelizumab + chemotherapy (PD-L1 CPS ≥ 10) (Active Comparator): Participants with a PD-L1 CPS ≥ 10 will receive after randomization placebo + tislelizumab + chemotherapy. The choice of one of three chemotherapy options is at the discretion of the investigator provided that it is either: (1) paclitaxel, (2) nab-paclitaxel, or (3) gemcitabine plus carboplatin.
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Placebo; Drug: Gemcitabine
- Arm D: ociperlimab + tislelizumab + chemotherapy (PD-L1 CPS score ≥ 1 to < 10) (Other): Exploratory arm: Participants with a PD-L1 CPS ≥ 1 to < 10 will receive ociperlimab + tislelizumab + chemotherapy. The choice of one of three chemotherapy options is at the discretion of the investigator provided that it is either: (1) paclitaxel, (2) nab-paclitaxel, or (3) gemcitabine plus carboplatin.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ociperlimab — 900 mg intravenously (IV) every 3 weeks (Q3W)
  Other Names: WCD118
  Arms: Arm A: ociperlimab+tislelizumab+chemotherapy (PD-L1 CPS ≥ 10); Arm D: ociperlimab + tislelizumab + chemotherapy (PD-L1 CPS score ≥ 1 to < 10)
Drug: Tislelizumab — 200 mg intravenously (IV) Q3W
  Other Names: VDT482
  Arms: Arm A: ociperlimab+tislelizumab+chemotherapy (PD-L1 CPS ≥ 10); Arm C: placebo + tislelizumab + chemotherapy (PD-L1 CPS ≥ 10); Arm D: ociperlimab + tislelizumab + chemotherapy (PD-L1 CPS score ≥ 1 to < 10)
Drug: Paclitaxel — 90 mg/m2 intravenously (IV) on Days 1, 8 and 15 every 28 days
Drug: Nab-paclitaxel — 100 mg/m2 intravenously (IV) on Days 1, 8 and 15 every 28 days
Drug: Carboplatin — AUC 2 intravenously (IV) on Days 1 and 8 every 21 days
Drug: Placebo — normal saline intravenously (IV) Q3W
  Arms: Arm B: placebo + pembrolizumab + chemotherapy (PD-L1 CPS ≥ 10); Arm C: placebo + tislelizumab + chemotherapy (PD-L1 CPS ≥ 10)
Drug: Pembrolizumab — 200 mg intravenously (IV) Q3W
  Other Names: MK-3475
  Arms: Arm B: placebo + pembrolizumab + chemotherapy (PD-L1 CPS ≥ 10)
Drug: Gemcitabine — 1000 mg/m2 intravenously (IV) on Days 1 and 8 every 21 days

SUMMARY:
The primary scientific question of interest of this study is whether the combination of ociperlimab, tislelizumab and chemotherapy improves progression-free survival (PFS) compared to the combination of placebo, pembrolizumab and chemotherapy as first-line therapy for adult men and women with advanced triple negative breast cancer (TNBC) whose tumors express programmed death ligand 1 (PD - L1) [combined positive score (CPS) ≥10], regardless of study treatment discontinuation or start of new anti-neoplastic therapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, Phase II study evaluating the efficacy and safety of ociperlimab in combination with tislelizumab and chemotherapy as first-line treatment for participants with advanced TNBC whose tumors express PD-L1 (CPS ≥ 10).

Additionally, the efficacy and safety of the triple combination (ociperlimab + tislelizumab + chemotherapy) will be assessed in Arm D (a separate single-arm, open-label cohort) in 30 participants with advanced TNBC whose tumors express PD-L1 (CPS ≥ 1 to < 10).

Study treatment will continue until the participant experiences one of the following: disease progression per investigator's assessment by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, unacceptable toxicity, pregnancy, treatment is discontinued at the discretion of the investigator or participant, start of a new antineoplastic therapy, withdrawal of consent, lost to follow-up, death, or study is terminated by the sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has histologically confirmed diagnosis of advanced (loco-regionally recurrent and not amenable to curative therapy, or metastatic (stage IV)) TNBC
* Participant has completed systemic treatment for Stage I-III breast cancer, if indicated, and ≥ 6 months have elapsed between the completion of systemic treatment with curative intent and disease recurrence
* A recently or newly obtained tumor biopsy from a metastatic site must be provided for determination of PD-L1 expression using the PD-L1 IHC 22C3 assay by a Novartis designated central laboratory, prior to study randomization. If a result of PD-L1 expression assessed by a PD-L1 IHC 22C3 pharmDx test in a local laboratory is available, this can serve as PD-L1 status confirmation. For Arms A, B and C participants must have PD-L1 positive tumors with CPS≥ 10. For Arm D, participants must have PD-L1 positive tumors with CPS ≥ 1 to < 10.
* Participant has measurable disease, i.e., at least one measurable lesion per RECIST 1.1 criteria (a lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation)
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participant has life expectancy ≥ 12 weeks from the start of study treatment

Key Exclusion Criteria:

* Participant has received prior treatment with immunotherapy in the metastatic setting, or anti-T cell immunoreceptor with Ig and ITIM domains (TIGIT) therapy in any setting
* History of severe hypersensitivity to any of the study drugs (i.e. monoclonal antibodies, gemcitabine, carboplatin, nab-paclitaxel, paclitaxel) or its excipients or to drugs of similar chemical classes
* Participant with inflammatory breast cancer at screening
* Participant has central nervous system (CNS) involvement which was not previously treated and/or was newly detected at screening. Previously treated CNS involvement must fulfill the following criteria to be eligible for the trial:

  1. Completed prior therapy (including radiation and/or surgery) for CNS metastases ≥ 28 days prior to the start of the study and
  2. CNS tumor is clinically stable at the time of screening, and
  3. Participant is not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases
* Participant has an active autoimmune diseases or history of autoimmune diseases that may relapse
* Participant has not recovered from all toxicities related to prior anticancer therapies to National Cancer Institute (NCI) CTCAE version 5.0 Grade ≤1. Exception to this criterion: participants with any grade of alopecia are allowed to enter the study

Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2029-07-17 (Estimated); Study Completion 2029-07-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) based on investigator assessment using RECIST 1.1 criteria in Arm A and B | From randomization to date of disease progression or death, assessed up to approximately 32 months after first randomization
  PFS is defined as the time from the date of randomization to the date of first documented progression or death due to any cause. The comparison of PFS between Arm A and Arm B will be provided

SECONDARY OUTCOMES:
Overall Survival (OS) based on investigator assessment using RECIST 1.1 criteria in Arm A, B and C | From randomization to death, assessed up to approximately 32 months after first randomization
  OS is defined as the time from date of randomization to date of death due to any cause. The comparison of OS between Arm A and Arm B, Arm B and Arm C, and Arm A and Arm C will be provided.
Overall Response Rate (ORR) based on investigator assessment using RECIST 1.1 criteria in Arm A, B and C | Up to approximately 32 months after first randomization
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) as per local assessment according to RECIST 1.1.
Clinical benefit rate (CBR) with confirmed response in Arm A, B and C | Approximately 32 months after first randomization
  CBR is defined as the percentage of participants with a BOR of confirmed CR, PR or stable disease (SD) lasting for a duration of 24 weeks. CR, PR and SD are defined as per local investigator assessment according to RECIST 1.1
Time to response (TTR) based on investigator assessment using RECIST 1.1 criteria in Arm A, B and C | From randomization to first documented response, assessed up to approximately 32 months after first randomization
  TTR is defined as the time from date of randomization to the first documented response of either CR or PR, as per local investigator assessment according to RECIST 1.1
Duration of Response (DOR) based on investigator assessment using RECIST 1.1 criteria in Arm A, B and C | From first documented response to disease progression or death, assessed up to approximately 32 months after first randomization
  DOR is defined as the duration of time between the date of first documented response (CR or PR as per local investigator assessment according to RECIST 1.1) and the date of first documented progression or death due to any cause.
Progression-free Survival (PFS) based on investigator assessment using RECIST 1.1 criteria in Arm A, B and C | From randomization to date of disease progression or death, assessed up to approximately 32 months after first randomization
  PFS is defined as the time from the date of randomization to the date of first documented progression or death due to any cause. PFS for participants in Arm C will be compared to PFS for participants in Arm A and B.
Number of participants with dose modifications | Approximately 32 months after first dose
  Number of participants with dose interruption and reductions for each drug component as a measure of tolerability
Anti-drug Antibodies (ADA) prevalence at Baseline for ociperlimab | Baseline
  prevalence at baseline is calculated as the percentage of participants who had an ADA positive result at baseline for ociperlimab
Anti-drug Antibodies (ADA) prevalence at Baseline for tislelizumab | Baseline
  prevalence at baseline is calculated as the percentage of participants who had an ADA positive result at baseline for tislelizumab
Anti-drug Antibodies (ADA) incidence on treatment for ociperlimab | From Cycle 1 to Cycle 16, end of treatment and 30 day safety follow-up. Each cycle is 21 days
  ADA incidence on treatment will be calculated as the percentage of participants who are treatment-induced ADA positive for ociperlimab
Anti-drug Antibodies (ADA) incidence on treatment for tislelizumab | From Cycle 1 to Cycle 16, end of treatment and 30 day safety follow-up. Each cycle is 21 days
  ADA incidence on treatment will be calculated as the percentage of participants who are treatment-induced ADA positive for tislelizumab
Change from baseline in the Functional Assessment of Cancer Therapy-Breast (FACT-B) Trial Outcomes Index (TOI) score | Up to approximately 32 months after first dose
  Change from baseline in the FACT-B TOI score for participants in Arms A, B and C. The FACT-B is a questionnaire that consists of 37 items with items from FACT-General (FACT-G) questionnaire (27 items) and from the Breast Cancer Subscale (BCS, 10 items). FACT-B consists of five subscales that address different aspects of the participant's quality of life: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and BCS. The FACT-B TOI is a composite of PWB, FWB and BCS, and ranges from 0 to 96, with higher scores indicating better quality of life.
Time to 5-point definitive deterioration in FACT-B TOI score | Up to approximately 32 months after first dose
  Time to 5-point definitive deterioration in the FACT-B TOI in Arms A, B and C. The FACT-B is a questionnaire that consists of 37 items with items from FACT-General (FACT-G) questionnaire (27 items) and from the Breast Cancer Subscale (BCS, 10 items). FACT-B consists of five subscales that address different aspects of the participant's quality of life: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and BCS. The FACT-B TOI is a composite of PWB, FWB and BCS, and ranges from 0 to 96, with higher scores indicating better quality of life. Definitive deterioration is defined as the time from the date of randomization to the date of event defined at least 5-point worsening from baseline with no later improvement above this threshold during the course of treatment or until death due to any cause, in the FACT-B TOI score.
Serum concentrations of ociperlimab | Cycle (C) 1 Day (D) 1, C1D2, C1D4, C1D8, C1D15, D1 of C2, C3, C4 and C5, C5D8, D1 of C6, C8, C12 and C16, end of treatment and 30 day post-treatment. Each cycle is 21 days.
  Summary statistics of serum ociperlimab concentrations by time point
Serum concentrations of tislelizumab | Cycle (C) 1 Day (D) 1, C1D2, C1D4, C1D8, C1D15, D1 of C2, C3, C4 and C5, C5D8, D1 of C6, C8, C12 and C16, end of treatment and 30 day post-treatment. Each cycle is 21 days.
  Summary statistics of serum tislelizumab concentrations by time point

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com